CLINICAL TRIAL: NCT00988754
Title: School Children and Adolescents as Health Experts - Step 3
Brief Title: School Based Health Promotion Program in Secondary Schools
Acronym: JuvenTUM 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Bavarian State Ministry of Health and Care (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LP00001 FA 08 07-26
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Cardiovascular Risk
Keywords: Obesity; childhood and adolescence; school and family-based lifestyle intervention; cardiovascular risk; Obesity and associated cardiovascular risk in childhood and adolescence,; health behaviour
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Medical examination once per year, school and family-based lifestyle intervention including a weekly health lesson, school-affiliation to sports clubs and regularly trainings for teachers and parents
  Interventions: Behavioral: School children and adolescents as health experts
- B (No Intervention): Medical examination and information on a healthy lifestyle.

INTERVENTIONS:
Behavioral: School children and adolescents as health experts — Experimental group: Weekly health lesson for children; Monthly training for teacher; 2-3 trainings/year for the parents
  Arms: A

SUMMARY:
The purpose of the study is to determine whether a school based health promotion program in secondary schools is effective with respect to an increase of physical activity, physical fitness and health.

DETAILED DESCRIPTION:
Current understanding of physical activity in childhood demonstrates the health benefits of regular exercise, such as improved cardiovascular fitness, skeletal health and prevention of overweight and obesity. The children obtained weekly health education lessons from their teachers to increase the physical activity in and outside of school and to improve health behavior (healthy food, no drugs) as well as the general well-being of children.

Monthly training for teachers and regular training (2-3x/year) for the parents complete the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children in the 1. grade of secondary General Schools or Intermediate Schools with written consent from the parents in the greater Munich area

Exclusion Criteria:

* Children without written consent from their parents

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 595 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Daily physical activity > 60 minutes | 4 years
  number of days with physical activity > 60 minutes

SECONDARY OUTCOMES:
Physical fitness | 4 years
  6-item-test battery (points)
Anthropometric parameters | 4 years
  BMI (kg/m2), BMI-SDS, Waist and upper arm circumferences (cm), skinfold thickness (mm), Blood pressure (mm Hg)
Blood samples | 4 years
  HDL-cholesterol (mg/dl), LDL-cholesterol (mg/dl), Triglycerides (mg/dl), Glucose (mg/dl), Insulin (µU/ml), Leptin (ng/ml), Adiponectin (µg/ml), Il-6 (pg/ml), hsCRP (mg/L)
Retinal vascular caliber | 4 years
  Central retinal arteriolar (CRAE) and venular (CRVE) vessel diameters, arteriolar-to-venular-ratio
Lifestyle and socio-economic index | 4 years
  Questionnaire concerning eating pattern, sitting behavior, smoking, drinking, school level parents, nationality children and parents)
Arterial stiffness | 4 years
  Sphygmograph
Quality of life | 4 years
  Questionnaire (KINDL-R)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Halle, Prof., M.D., Study Chair — Department of Medicine, Division of Prevention, Rehabilitation and Sports Medicine, Technical University Munich, Germany
Locations (1):
- Department of Medicine, Division of Prevention, Rehabilitation and Sports Medicine, Technical University Munich, Munich, Bavaria, Germany

REFERENCES:
- [Background] Baker JL, Olsen LW, Sorensen TI. Childhood body-mass index and the risk of coronary heart disease in adulthood. N Engl J Med. 2007 Dec 6;357(23):2329-37. doi: 10.1056/NEJMoa072515. PMID 18057335
- [Background] Bibbins-Domingo K, Coxson P, Pletcher MJ, Lightwood J, Goldman L. Adolescent overweight and future adult coronary heart disease. N Engl J Med. 2007 Dec 6;357(23):2371-9. doi: 10.1056/NEJMsa073166. PMID 18057339
- [Background] Owen CG, Whincup PH, Orfei L, Chou QA, Rudnicka AR, Wathern AK, Kaye SJ, Eriksson JG, Osmond C, Cook DG. Is body mass index before middle age related to coronary heart disease risk in later life? Evidence from observational studies. Int J Obes (Lond). 2009 Aug;33(8):866-77. doi: 10.1038/ijo.2009.102. Epub 2009 Jun 9. PMID 19506565
- [Background] Birch LL, Ventura AK. Preventing childhood obesity: what works? Int J Obes (Lond). 2009 Apr;33 Suppl 1:S74-81. doi: 10.1038/ijo.2009.22. PMID 19363514
- [Background] Saarelainen H, Valtonen P, Punnonen K, Laitinen T, Raitakari OT, Juonala M, Heiskanen N, Lyyra-Laitinen T, Viikari JS, Heinonen S. Flow mediated vasodilation and circulating concentrations of high sensitive C-reactive protein, interleukin-6 and tumor necrosis factor-alpha in normal pregnancy--The Cardiovascular Risk in Young Finns Study. Clin Physiol Funct Imaging. 2009 Sep;29(5):347-52. doi: 10.1111/j.1475-097X.2009.00877.x. Epub 2009 Jun 1. PMID 19489963
- [Background] Magnussen CG, Venn A, Thomson R, Juonala M, Srinivasan SR, Viikari JS, Berenson GS, Dwyer T, Raitakari OT. The association of pediatric low- and high-density lipoprotein cholesterol dyslipidemia classifications and change in dyslipidemia status with carotid intima-media thickness in adulthood evidence from the cardiovascular risk in Young Finns study, the Bogalusa Heart study, and the CDAH (Childhood Determinants of Adult Health) study. J Am Coll Cardiol. 2009 Mar 10;53(10):860-9. doi: 10.1016/j.jacc.2008.09.061. PMID 19264243
- [Background] Harris KC, Kuramoto LK, Schulzer M, Retallack JE. Effect of school-based physical activity interventions on body mass index in children: a meta-analysis. CMAJ. 2009 Mar 31;180(7):719-26. doi: 10.1503/cmaj.080966. PMID 19332753
- [Background] Daniels SR, Arnett DK, Eckel RH, Gidding SS, Hayman LL, Kumanyika S, Robinson TN, Scott BJ, St Jeor S, Williams CL. Overweight in children and adolescents: pathophysiology, consequences, prevention, and treatment. Circulation. 2005 Apr 19;111(15):1999-2012. doi: 10.1161/01.CIR.0000161369.71722.10. PMID 15837955
- [Background] Hayman LL, Williams CL, Daniels SR, Steinberger J, Paridon S, Dennison BA, McCrindle BW; Committee on Atherosclerosis, Hypertension, and Obesity in Youth (AHOY) of the Council on Cardiovascular Disease in the Young, American Heart Association. Cardiovascular health promotion in the schools: a statement for health and education professionals and child health advocates from the Committee on Atherosclerosis, Hypertension, and Obesity in Youth (AHOY) of the Council on Cardiovascular Disease in the Young, American Heart Association. Circulation. 2004 Oct 12;110(15):2266-75. doi: 10.1161/01.CIR.0000141117.85384.64. No abstract available. PMID 15477426
- [Background] McCall A, Raj R. Exercise for prevention of obesity and diabetes in children and adolescents. Clin Sports Med. 2009 Jul;28(3):393-421. doi: 10.1016/j.csm.2009.03.001. PMID 19505623
- [Background] Oetzel KB, Scott AA, McGrath J. School-based health centers and obesity prevention: changing practice through quality improvement. Pediatrics. 2009 Jun;123 Suppl 5:S267-71. doi: 10.1542/peds.2008-2780D. PMID 19470602
- [Background] Dunford LJ, Langley-Evans SC, McMullen S. Childhood obesity and adult cardiovascular disease risk: a systematic review. Int J Obes (Lond). 2010 Jan;34(1):18-28. doi: 10.1038/ijo.2009.61. Epub 2009 May 12. PMID 19434067
- [Background] Bruss MB, Michael TJ, Morris JR, Applegate B, Dannison L, Quitugua JA, Palacios RT, Klein DJ. Childhood obesity prevention: an intervention targeting primary caregivers of school children. Obesity (Silver Spring). 2010 Jan;18(1):99-107. doi: 10.1038/oby.2009.111. Epub 2009 May 7. PMID 19424164
- [Derived] Siegrist M, Heitkamp M, Braun I, Vogg N, Haller B, Langhof H, Koenig W, Halle M. Changes of omentin-1 and chemerin during 4 weeks of lifestyle intervention and 1 year follow-up in children with obesity. Clin Nutr. 2021 Nov;40(11):5648-5654. doi: 10.1016/j.clnu.2021.09.042. Epub 2021 Oct 8. PMID 34666255
- [Derived] Siegrist M, Hanssen H, Lammel C, Haller B, Koch AM, Stemp P, Dandl E, Liestak R, Parhofer KG, Vogeser M, Halle M. Effects of a cluster-randomized school-based prevention program on physical activity and microvascular function (JuvenTUM 3). Atherosclerosis. 2018 Nov;278:73-81. doi: 10.1016/j.atherosclerosis.2018.09.003. Epub 2018 Sep 8. PMID 30261471
- [Derived] Hanssen H, Siegrist M, Neidig M, Renner A, Birzele P, Siclovan A, Blume K, Lammel C, Haller B, Schmidt-Trucksass A, Halle M. Retinal vessel diameter, obesity and metabolic risk factors in school children (JuvenTUM 3). Atherosclerosis. 2012 Mar;221(1):242-8. doi: 10.1016/j.atherosclerosis.2011.12.029. Epub 2011 Dec 27. PMID 22244041
- [Derived] Siegrist M, Hanssen H, Lammel C, Haller B, Halle M. A cluster randomised school-based lifestyle intervention programme for the prevention of childhood obesity and related early cardiovascular disease (JuvenTUM 3). BMC Public Health. 2011 Apr 22;11:258. doi: 10.1186/1471-2458-11-258. PMID 21513530
- See also: Related Info — http://www.juventum.med.tum.de